CLINICAL TRIAL: NCT02177760
Title: Sirolimus in Prevention of aGVHD in Maternally Engrafted (TME) Severe Combined Immunodeficiency (SCID) Infants Receiving Unconditioned Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Sirolimus Prophylaxis for aGVHD in TME SCID
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Preliminary data suggested a better approach available
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-13024
Record Dates: First submitted 2014-06-19; First posted 2014-06-30 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Severe Combined Immunodeficiency; Transplacental Maternal Engraftment; Stem Cell Transplant
Keywords: SCID; severe combined immunodeficiency; maternal engraftment; aGVHD prophylaxis; sirolimus
MeSH Terms: conditions — Severe Combined Immunodeficiency | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): Sirolimus (0.05 mg/kg/day) day -5 for aGVHD prophylaxis through day +100 or until T-regulatory cells >9% of CD4 effector cells; whichever comes first.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus
  Other Names: Rapamune

SUMMARY:
Study Design: SCID infants receiving an unconditioned haploidentical transplant will be started on Sirolimus (0.05 mg/kg/day) day -5 for Acute Graft-Versus-Host Disease (aGVHD) prophylaxis. Sirolimus levels will be monitored with goal sirolimus trough level of 5-8 ng/mL. Patients will be monitored for signs of aGVHD as defined by UCSF SOP CL 221.06 through day +100. Sirolimus will be tapered once T-regulatory cell to CD4 effector cell ratio is > or = 9%.

Setting: Inpatient BMT Unit Benioff Children's Hospital at UCSF Medical Center

Study Subjects: 15 infants with diagnosis of maternally engrafted T cells SCID by CA Newborn screen receiving unconditioned haploidentical HSCT

Main Outcome Measures: Incidence of aGVHD (dermatitis, hepatitis, enteritis) as defined by SOP CL 221.06 by Day +100.

Hypothesis 1. Patients placed on sirolimus prophylaxis will have lower incidence of aGVHD compared to historical controls.

Hypothesis 2. Lower doses of sirolimus milligram per kilogram will be required to maintain goal troughs of 5-8 ng/mL.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with SCID on CA newborn screen
* Evidence of Maternal Engraftment
* Unconditioned haploidentical hematopoeitic stem cell transplant

Exclusion Criteria:

* Evidence of acute graft vs. host disease

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Incidence of aGVHD | 105 days
  Incidence of aGVHD (dermatitis, hepatitis, enteritis) as defined by UCSF SOP CL 221.06 by Day +100.

SECONDARY OUTCOMES:
T-regulatory cell enumeration | 105 days
  T-regulatory cell enumeration studies by blood draw prior to prophylaxis and at day +30, day+60, day+100.
Sirolimus therapeutic drug monitoring | 105 days
  Sirolimus therapeutic drug monitoring will be done via blood draws(after initial 4th dose; thereafter every 4th dose with adjustment; once stable it will be measured weekly). We will determine the average dose in milligrams per kilograms that would be needed to reach therapeutic trough levels of 5-8 ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Dvorak, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Benioff Children's Hospital at UCSF Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Buckley RH, Schiff SE, Schiff RI, Markert L, Williams LW, Roberts JL, Myers LA, Ward FE. Hematopoietic stem-cell transplantation for the treatment of severe combined immunodeficiency. N Engl J Med. 1999 Feb 18;340(7):508-16. doi: 10.1056/NEJM199902183400703. PMID 10021471
- [Background] Dvorak CC, Cowan MJ. Hematopoietic stem cell transplantation for primary immunodeficiency disease. Bone Marrow Transplant. 2008 Jan;41(2):119-26. doi: 10.1038/sj.bmt.1705890. Epub 2007 Oct 29. PMID 17968328
- [Background] Muller SM, Ege M, Pottharst A, Schulz AS, Schwarz K, Friedrich W. Transplacentally acquired maternal T lymphocytes in severe combined immunodeficiency: a study of 121 patients. Blood. 2001 Sep 15;98(6):1847-51. doi: 10.1182/blood.v98.6.1847. PMID 11535520
- [Background] Pulsipher MA, Wall DA, Grimley M, Goyal RK, Boucher KM, Hankins P, Grupp SA, Bunin N. A phase I/II study of the safety and efficacy of the addition of sirolimus to tacrolimus/methotrexate graft versus host disease prophylaxis after allogeneic haematopoietic cell transplantation in paediatric acute lymphoblastic leukaemia (ALL). Br J Haematol. 2009 Dec;147(5):691-9. doi: 10.1111/j.1365-2141.2009.07889.x. Epub 2009 Sep 10. PMID 19744131
- [Background] Cutler C, Antin JH. Sirolimus immunosuppression for graft-versus-host disease prophylaxis and therapy: an update. Curr Opin Hematol. 2010 Nov;17(6):500-4. doi: 10.1097/MOH.0b013e32833e5b2e. PMID 20717025
- [Background] Pulsipher MA, Langholz B, Wall DA, Schultz KR, Bunin N, Carroll WL, Raetz E, Gardner S, Gastier-Foster JM, Howrie D, Goyal RK, Douglas JG, Borowitz M, Barnes Y, Teachey DT, Taylor C, Grupp SA. The addition of sirolimus to tacrolimus/methotrexate GVHD prophylaxis in children with ALL: a phase 3 Children's Oncology Group/Pediatric Blood and Marrow Transplant Consortium trial. Blood. 2014 Mar 27;123(13):2017-25. doi: 10.1182/blood-2013-10-534297. Epub 2014 Feb 4. PMID 24497539
- [Background] Yong PL, Russo P, Sullivan KE. Use of sirolimus in IPEX and IPEX-like children. J Clin Immunol. 2008 Sep;28(5):581-7. doi: 10.1007/s10875-008-9196-1. Epub 2008 May 15. PMID 18481161
- [Background] Strauss L, Czystowska M, Szajnik M, Mandapathil M, Whiteside TL. Differential responses of human regulatory T cells (Treg) and effector T cells to rapamycin. PLoS One. 2009 Jun 22;4(6):e5994. doi: 10.1371/journal.pone.0005994. PMID 19543393
- [Background] Fujioka T, Tamaki H, Ikegame K, Yoshihara S, Taniguchi K, Kaida K, Kato R, Inoue T, Nakata J, Ishii S, Soma T, Okada M, Ogawa H. Frequency of CD4(+)FOXP3(+) regulatory T-cells at early stages after HLA-mismatched allogeneic hematopoietic SCT predicts the incidence of acute GVHD. Bone Marrow Transplant. 2013 Jun;48(6):859-64. doi: 10.1038/bmt.2012.232. Epub 2012 Nov 19. PMID 23165499